CLINICAL TRIAL: NCT04234399
Title: Determination of the Diagnostic Detection Rate of Axumin (Fluciclovine) PET/CT Utilizing the High Resolution Digital Philips Vereos Scanner, in Patients With Biochemical Recurrence After Radical Prostatectomy
Brief Title: Determination of the Diagnostic Detection Rate of Axumin (Fluciclovine) Digital PET/CT, Post-prostatectomy
Status: Terminated | Type: Observational
Why Stopped: Lack of efficacy of Axumin and resultant lack of interest in recruitment. FDA approval of PSMA also hampered enrollment.
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Dmitriy Akselrod, MD, Assistant Professor, University of Vermont
Other Study IDs: UVMCC1905; BED-IIT 280 (Other Grant/Funding Number: Blue Earth Diagnostics)
Record Dates: First submitted 2020-01-14; First posted 2020-01-21 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Prostatic Neoplasm
Keywords: Recurrence; Fluciclovine; Axumin; PSA
MeSH Terms: conditions — Prostatic Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Group: All patients receiving SOC imaging and Axumin PET scans.
  Interventions: Diagnostic Test: Fluciclovine PET/CT using a digital PET/CT

INTERVENTIONS:
Diagnostic Test: Fluciclovine PET/CT using a digital PET/CT — Fluciclovine is a radiotracer that will be used in conjunction with the high resolution digital Vereos PET/CT scanner.

SUMMARY:
Fluciclovine F18 (Axumin) has been demonstrated to provide good delineation of recurrence of prostate cancer after definitive therapies. Fluciclovine in conjunction with the high-resolution digital Vereos (Phillips) PET-CT scanner may detect low volume recurrence in the prostatectomy bed or metastatic site (s).

20-40 % of men will suffer a biochemical recurrence of their prostate cancer after radical prostatectomy, depending on their final pathological staging, defined as a rising PSA > 0.2 ng/ml.

The ability to more accurately diagnose local recurrence (i.e. pelvis) or oligometastasis may lead to the opportunity of precise therapy of these sites with more durable cancer responses, less morbidity and potential cure in selective men after Radical Prostatectomy.

The ability to diagnose widespread metastatic Prostate Cancer after Radical Prostatectomy, or disease that is inaccessible to local selective therapies would spare these men the cost and morbidity of inappropriate therapy.

The diagnosis of true stage D0 Prostate Cancer (No objective evidence of metastases) in men after Radical Prostatectomy would yield improved overall and disease specific survival if Androgen Deprivation Therapy was initiated at its earliest stage. This would also obviate the need for inappropriate local therapies (i.e. pelvic radiotherapy).

The aim is to compare the detection rate of standard of care (CT Pelvis/Abdomen, MR Pelvis, Bone Scan) with Fluciclovine PET/CT performed on the Vereos Philips Scanner. The study aims to compare the performance of Digital (high resolution) PET to CT/MRI/Bone scan rather than analog (lower resolution) PET. Prior studies have tested analog PET compared to other modalities. One could make an inference that if our study's Digital PET performs better than the performance of Analog PET in those studies, then Digital PET should have a better detection rate than Analog PET. However, investigators are not making a direct comparison between digital and Analog in our comparison.

DETAILED DESCRIPTION:
Aim:

Compare the detection rate of standard of care (CT Pelvis/Abdomen, MR Pelvis, Bone Scan) with Fluciclovine PET/CT performed on the Vereos Philips Scanner. The study aims to compare the performance of Digital (high resolution) PET to CT/MRI/Bone scan rather than analog (lower resolution) PET. This was reported in Michopoulou S, O'Shaughnessy E, Thomson K, Guy MJ. Discovery Molecular Imaging Digital Ready PET/CT performance evaluation according to the NEMA NU2-2012 standard. Nucl Med Commun. 2018 Nov 27; doi:10.1097/MNM.0000000000000962. Prior studies have tested analog PET compared to other modalities. One could make an inference that if our study's Digital PET performs better than the performance of Analog PET in those studies, then Digital PET should have a better detection rate than Analog PET. However, investigators are not making a direct comparison between digital and Analog in our comparison.

Background:

Fluciclovine F18 (Fluciclovine) has been demonstrated to provide good delineation of recurrence of prostate cancer after definitive therapies (Odewole OA et al 2016). Fluciclovine in conjunction with the high-resolution digital Vereos (Phillips) PET-CT scanner may detect low volume recurrence in the prostatectomy bed or metastatic site (s).

20-40 % of men will suffer a biochemical recurrence of their prostate cancer after radical prostatectomy, depending on their final pathological staging, defined as a rising PSA > 0.2 ng/ml.

The ability to more accurately diagnose local recurrence (i.e. pelvis) or oligometastasis may lead to the opportunity of precise therapy of these sites with more durable cancer responses, less morbidity and potential cure in selective men after Radical Prostatectomy.

The ability to diagnose widespread metastatic Prostate Cancer after Radical Prostatectomy, or disease that is inaccessible to local selective therapies would spare these men the cost and morbidity of inappropriate therapy.

The diagnosis of true stage D0 Prostate Cancer (No objective evidence of metastases) in men after Radical Prostatectomy would yield improved overall and disease specific survival if Androgen Deprivation Therapy was initiated at its earliest stage. This would also obviate the need for inappropriate local therapies (i.e. pelvic radiotherapy).

Preliminary Studies:

The safety, efficacy, reproducibility, and reliability of Fluciclovine was initially evaluated by the Emory group in men with suspected recurrence of prostate cancer based on rising PSA levels following radical prostatectomy and/or radiotherapy. Fluciclovine's safety, detection rate, and diagnostic performance was further validated in a multi-site data aggregation study using data from Emory, Noway, and Italy.

The performance of Fluciclovine seems to be affected by degree of PSA elevation. Statistically significant difference in performance compared to CT was found at PSA levels >1 ng/ml. However, at a PSA level of <1 ng/ml, no statistically significant difference was found by Odewole et al. These findings were independent of PSA doubling time and Gleason Score.

The Bologna study evaluated the concordance between Fluciclovine and C11 Choline scans in patients with median PSA value of 1.44 ng/ml (interquartile range = 0.78 to 2.8 ng/ml).5 The accuracy of Fluciclovine was 38% vs 32% for C11 Choline. In a subsequent Emory study which studied Fluciclovine without a correlative imaging test, Fluciclovine scan detected recurrence in 72% (18/25) of patients with PSA of <1 ng/ml. However, there was no reconciliation of false positive examinations, as all abnormal radiotracer uptake were deemed a true positive. Performance of Fluciclovine was again noted to improve with increasing PSA levels, at 83% (5/6) for PSA of 1-<2 ng/ml and 100% (11/11) for PSA>= 2 ng/ml.

Rationale:

A Fluciclovine scan can detect and localize recurrent prostate cancer. Fluciclovine is an FDA-approved diagnostic imaging agent, also known as a "tracer," which may help determine if and where the prostate cancer has recurred.

Procedures:

Fluciclovine is used as a tracer for a PET/CT scan. Patients will need to prepare for the Fluciclovine (fluciclovine F 18) injection and scan. They will need avoid any significant exercise for at least a full 24 hours prior to Fluciclovine PET/CT scan and not eat or drink for at least 4 hours prior to PET/CT scan (other than small amounts of water for taking medications).

With respect to determining if a finding is true positive, investigators will follow the following process. The research PET scan of each patient and SOC imaging will be read by radiologists blinded to the results of the other test. The results of both will then be reviewed by PI for concordance. If the research PET scan finds sites of disease that were not identified on SOC imaging, the case will be brought to Interdisciplinary UVMMC Genitourinary tumor board. Depending on the site of disease and presence of other concordant sites of metastatic disease between scans, it may have no impact on the SOC treatment. If it is deemed by the UVMMC Genitourinary Tumor Board that it will have a meaningful impact on treatment decisions and the detected lesion is accessible to be safely sampled, the patient will be approached by their treating physician to discuss the discordant findings, their significance, and the rationale behind a biopsy and its impact on their care.

The sampling will then be performed a part of standard-of-care work-up, given that these patients would have been eligible for Fluciclovine PET imaging in this setting, per FDA label. Given the low PSA range of our target population in this study, the likelihood that these lesions would be amenable to sampling using conventional image guidance is low. Therefore, in cases where the research scan finds additional disease that would alter therapy, the decision of whether to act on it will be based on the overall clinical scenario of each patient, and will be decided by the treating team with the support of the UVMMC Genitourinary Tumor Board.

ELIGIBILITY:
Inclusion Criteria:

1. Prostatectomy patients with previously undetectable PSA and subsequent biochemical recurrence defined by PSA between 0.2 ng/ml and 1.0 ng/ml within 90 days prior to Fluciclovine scan
2. Age >40
3. Ability to provide informed consent

Exclusion Criteria:

1. History of allergic reaction to Fluciclovine
2. Anti Androgen treatment in the 6 months prior to enrollment
3. Any patient whose body habitus, as determined by radiology personnel, will effectively inhibit the ability to obtain PET/CT imaging or will interfere with the images so as to make them clinically uninterpretable.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prostatectomy patients with previously undetectable PSA and subsequent biochemical recurrence defined by PSA between 0.2 ng/ml and 1.0 ng/ml within 90 days prior to Fluciclovine scan
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Detection rate | Patients will be scheduled for both SOC imaging as well as the Fluciclovine PET within 4 weeks of screening and signing of informed consent. The detection rates between SOC and Fluciclovine scans will be compared.
  Comparison of Fluciclovine digital PET/CT with standard of care imaging. Single time point.

CONTACTS AND LOCATIONS:
Locations (1):
- UVM Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schuster DM, Nieh PT, Jani AB, Amzat R, Bowman FD, Halkar RK, Master VA, Nye JA, Odewole OA, Osunkoya AO, Savir-Baruch B, Alaei-Taleghani P, Goodman MM. Anti-3-[(18)F]FACBC positron emission tomography-computerized tomography and (111)In-capromab pendetide single photon emission computerized tomography-computerized tomography for recurrent prostate carcinoma: results of a prospective clinical trial. J Urol. 2014 May;191(5):1446-53. doi: 10.1016/j.juro.2013.10.065. Epub 2013 Oct 19. PMID 24144687
- [Background] Odewole OA, Oyenuga OA, Tade F, Savir-Baruch B, Nieh PT, Master V, Chen Z, Wang X, Jani AB, Bellamy LM, Halkar RK, Goodman MM, Schuster DM. Reproducibility and reliability of anti-3-[(1)(8)F]FACBC uptake measurements in background structures and malignant lesions on follow-up PET-CT in prostate carcinoma: an exploratory analysis. Mol Imaging Biol. 2015 Apr;17(2):277-83. doi: 10.1007/s11307-014-0797-1. PMID 25281411
- [Background] Schuster DM, Savir-Baruch B, Nieh PT, Master VA, Halkar RK, Rossi PJ, Lewis MM, Nye JA, Yu W, Bowman FD, Goodman MM. Detection of recurrent prostate carcinoma with anti-1-amino-3-18F-fluorocyclobutane-1-carboxylic acid PET/CT and 111In-capromab pendetide SPECT/CT. Radiology. 2011 Jun;259(3):852-61. doi: 10.1148/radiol.11102023. Epub 2011 Apr 14. PMID 21493787
- [Background] Odewole OA, Tade FI, Nieh PT, Savir-Baruch B, Jani AB, Master VA, Rossi PJ, Halkar RK, Osunkoya AO, Akin-Akintayo O, Zhang C, Chen Z, Goodman MM, Schuster DM. Recurrent prostate cancer detection with anti-3-[(18)F]FACBC PET/CT: comparison with CT. Eur J Nucl Med Mol Imaging. 2016 Sep;43(10):1773-83. doi: 10.1007/s00259-016-3383-8. Epub 2016 Apr 18. PMID 27091135
- [Background] Nanni C, Zanoni L, Pultrone C, Schiavina R, Brunocilla E, Lodi F, Malizia C, Ferrari M, Rigatti P, Fonti C, Martorana G, Fanti S. (18)F-FACBC (anti1-amino-3-(18)F-fluorocyclobutane-1-carboxylic acid) versus (11)C-choline PET/CT in prostate cancer relapse: results of a prospective trial. Eur J Nucl Med Mol Imaging. 2016 Aug;43(9):1601-10. doi: 10.1007/s00259-016-3329-1. Epub 2016 Mar 10. PMID 26960562
- [Background] Akin-Akintayo OO, Jani AB, Odewole O, Tade FI, Nieh PT, Master VA, Bellamy LM, Halkar RK, Zhang C, Chen Z, Goodman MM, Schuster DM. Change in Salvage Radiotherapy Management Based on Guidance With FACBC (Fluciclovine) PET/CT in Postprostatectomy Recurrent Prostate Cancer. Clin Nucl Med. 2017 Jan;42(1):e22-e28. doi: 10.1097/RLU.0000000000001379. PMID 27749412
- [Background] Bruce JY, Lang JM, McNeel DG, Liu G. Current controversies in the management of biochemical failure in prostate cancer. Clin Adv Hematol Oncol. 2012 Nov;10(11):716-22. PMID 23271258
- [Background] Paller CJ, Antonarakis ES. Management of biochemically recurrent prostate cancer after local therapy: evolving standards of care and new directions. Clin Adv Hematol Oncol. 2013 Jan;11(1):14-23. PMID 23416859
- [Background] Ost P, Reynders D, Decaestecker K, Fonteyne V, Lumen N, De Bruycker A, Lambert B, Delrue L, Bultijnck R, Claeys T, Goetghebeur E, Villeirs G, De Man K, Ameye F, Billiet I, Joniau S, Vanhaverbeke F, De Meerleer G. Surveillance or Metastasis-Directed Therapy for Oligometastatic Prostate Cancer Recurrence: A Prospective, Randomized, Multicenter Phase II Trial. J Clin Oncol. 2018 Feb 10;36(5):446-453. doi: 10.1200/JCO.2017.75.4853. Epub 2017 Dec 14. PMID 29240541
- [Background] Radwan N, Phillips R, Ross A, Rowe SP, Gorin MA, Antonarakis ES, Deville C, Greco S, Denmeade S, Paller C, Song DY, Diehn M, Wang H, Carducci M, Pienta KJ, Pomper MG, DeWeese TL, Dicker A, Eisenberger M, Tran PT. A phase II randomized trial of Observation versus stereotactic ablative RadiatIon for OLigometastatic prostate CancEr (ORIOLE). BMC Cancer. 2017 Jun 29;17(1):453. doi: 10.1186/s12885-017-3455-6. PMID 28662647
- [Background] Smith MR, Saad F, Chowdhury S, Oudard S, Hadaschik BA, Graff JN, Olmos D, Mainwaring PN, Lee JY, Uemura H, Lopez-Gitlitz A, Trudel GC, Espina BM, Shu Y, Park YC, Rackoff WR, Yu MK, Small EJ; SPARTAN Investigators. Apalutamide Treatment and Metastasis-free Survival in Prostate Cancer. N Engl J Med. 2018 Apr 12;378(15):1408-1418. doi: 10.1056/NEJMoa1715546. Epub 2018 Feb 8. PMID 29420164
- [Background] Bach-Gansmo T, Nanni C, Nieh PT, Zanoni L, Bogsrud TV, Sletten H, Korsan KA, Kieboom J, Tade FI, Odewole O, Chau A, Ward P, Goodman MM, Fanti S, Schuster DM, Willoch F. Multisite Experience of the Safety, Detection Rate and Diagnostic Performance of Fluciclovine (18F) Positron Emission Tomography/Computerized Tomography Imaging in the Staging of Biochemically Recurrent Prostate Cancer. J Urol. 2017 Mar;197(3 Pt 1):676-683. doi: 10.1016/j.juro.2016.09.117. Epub 2016 Oct 13. PMID 27746282
- [Background] Andriole GL, Kostakoglu L, Chau A, Duan F, Mahmood U, Mankoff DA, Schuster DM, Siegel BA; LOCATE Study Group. The Impact of Positron Emission Tomography with 18F-Fluciclovine on the Treatment of Biochemical Recurrence of Prostate Cancer: Results from the LOCATE Trial. J Urol. 2019 Feb;201(2):322-331. doi: 10.1016/j.juro.2018.08.050. PMID 30179618
- See also: Axumin FDA prescribing information — https://www.accessdata.fda.gov/drugsatfda_docs/label/2016/208054s000lbl.pdf